CLINICAL TRIAL: NCT02227940
Title: A Phase I Study of Ceritinib (LDK378), a Novel ALK Inhibitor, in Combination With Gemcitabine-Based Chemotherapy in Patients With Advanced Solid Tumors
Brief Title: Ceritinib and Combination Chemotherapy in Treating Patients With Advanced Solid Tumors or Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 248813; NCI-2014-01766 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 248813 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Advanced Malignant Solid Neoplasm; ALK Positive; Metastatic Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ceritinib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (ceritinib MTD then with gemcitabine alone) (Experimental): Dose Escalation Cohort 1: Patients with advanced solid tumors for whom gemcitabine hydrochloride-based therapy is clinically appropriate receive ceritinib PO (QD on days 1-28 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Expansion Cohort 1E: Once the MTD of ceritinib has been determined, an additional 10 patients with ALK-positive advanced solid tumors who previously progressed on gemcitabine hydrochloride-based therapy receive ceritinib and gemcitabine hydrochloride as in the dose escalation cohort 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ceritinib; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm 2 (ceritinib MTD then with gemcitabine and nab-paclitaxel) (Experimental): Dose Escalation Cohort 2: Patients with advanced pancreatic cancer receive ceritinib PO QD on days 1-28, gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15, and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Expansion Cohort 2E: Once the MTD of ceritinib has been determined, patients with ALK-positive advanced solid tumors receive ceritinib, gemcitabine hydrochloride, and paclitaxel albumin-stabilized nanoparticle formulation as in the dose escalation cohort 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ceritinib; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Other: Pharmacological Study
- Arm 3 (ceritinib MTD then with gemcitabine and cisplatin) (Experimental): Dose Escalation Cohort 3: Patients with advanced solid tumors for whom gemcitabine hydrochloride and cisplatin-based therapy is clinically appropriate receive ceritinib PO QD on days 1-28, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and cisplatin IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Expansion Cohort 3E: Once the MTD of ceritinib has been determined, an additional 10 patients with ALK-positive advanced solid tumors receive ceritinib, gemcitabine hydrochloride, and cisplatin as in the dose escalation cohort 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ceritinib; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Ceritinib — Given PO
  Other Names: LDK 378; LDK378; Zykadia
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm 3 (ceritinib MTD then with gemcitabine and cisplatin)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; nab-paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; protein-bound paclitaxel
  Arms: Arm 2 (ceritinib MTD then with gemcitabine and nab-paclitaxel)
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of ceritinib and combination chemotherapy in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or pancreatic cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or has spread to other places in the body (metastatic). Ceritinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, paclitaxel albumin-stabilized nanoparticle formulation, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ceritinib and more than one drug (combination chemotherapy) may be a better treatment for solid tumors or pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D) of ceritinib in combination with gemcitabine (gemcitabine hydrochloride) alone, gemcitabine/nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) and gemcitabine/cisplatin in patients with advanced solid malignancies.

SECONDARY OBJECTIVES:

I. Characterize the safety profile of ceritinib in combination with gemcitabine based chemotherapy in advanced solid malignancies.

II. Determine the pharmacokinetic profile of ceritinib, gemcitabine, nab-paclitaxel, cisplatin and their metabolites when administered in combination in patients with advanced solid tumors.

III. Determine the preliminary efficacy of the study combinations.

TERTIARY OBJECTIVES:

I. Explore potential biomarkers of efficacy to the study combination.

OUTLINE: This is a dose-escalation study of ceritinib. Patients are assigned to 1 of 3 treatment arms.

ARM 1 (ceritinib MTD then with gemcitabine alone):

Dose Escalation Cohort 1: Patients with advanced solid tumors for whom gemcitabine hydrochloride-based therapy is clinically appropriate receive ceritinib orally (PO) once daily (QD) on days 1-28 and gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Expansion Cohort 1E: Once the MTD of ceritinib has been determined, an additional 10 patients with anaplastic lymphoma kinase positive (ALK-positive) advanced solid tumors who previously progressed on gemcitabine hydrochloride-based therapy receive ceritinib and gemcitabine hydrochloride as in the dose escalation cohort 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 2 (ceritinib MTD then with gemcitabine and nab-paclitaxel):

Dose Escalation Cohort 2: Patients with advanced pancreatic cancer receive ceritinib PO QD on days 1-28, gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15, and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Expansion Cohort 2E: Once the MTD of ceritinib has been determined, patients with ALK-positive advanced solid tumors receive ceritinib, gemcitabine hydrochloride, and paclitaxel albumin-stabilized nanoparticle formulation as in the dose escalation cohort 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 3 (ceritinib MTD then with gemcitabine and cisplatin):

Dose Escalation Cohort 3: Patients with advanced solid tumors for whom gemcitabine hydrochloride and cisplatin-based therapy is clinically appropriate receive ceritinib PO QD on days 1-28, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and cisplatin IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Expansion Cohort 3E: Once the MTD of ceritinib has been determined, an additional 10 patients with ALK-positive advanced solid tumors receive ceritinib, gemcitabine hydrochloride, and cisplatin as in the dose escalation cohort 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1: histologically or cytologically confirmed solid tumors that are advanced that gemcitabine-based treatment is considered a clinically appropriate option
* Arm 2: histologically or cytologically confirmed adenocarcinoma of the pancreas that is locally advanced or metastatic
* Arm 3: histologically or cytologically confirmed solid tumors that are advanced that gemcitabine plus cisplatin treatment is considered a clinically appropriate option
* Arms 1E, 2E and 3E: solid tumor that demonstrate anaplastic lymphoma kinase (ALK) positivity; ALK positivity can be assessed using the assays below, and documentation of ALK positivity using one of the tests below is required

  * Fluorescence in situ hybridization (FISH) test for ALK positivity using the Food and Drug Administration (FDA)-approved FISH test (Abbott Molecular Inc), using Vysis breakapart probes (defined as 15% or more positive tumor cells); OR
  * Harboring a confirmed ALK positivity, as determined by positivity to the Ventana immunohistochemistry (IHC) assay
* Arms 1E: previously treated with and progressed on gemcitabine-containing therapy
* Arms 1, 2, 3: patients should have clinically measurable or evaluable malignant disease
* Arms 1E, 2E, 3E: patients with at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 that have not been previously irradiated
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy >= 3 months
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (system international [SI] units 1.5 x 10^9/L)
* Platelets >= 100,000 cells/mm^3 (SI units 100 x 10^9/L)
* Hemoglobin >= 9 g/dL (SI units 90 g/L) (in the absence of transfusion within 24 hours prior to dosing)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3 x upper limit of normal (ULN); in patients with known hepatic involvement, AST and ALT =< 5 x ULN are allowed
* Total bilirubin =< 1.5 x ULN
* Calculated or measured creatinine clearance (CrCL) >= 60 mL/min using modified Cockcroft and Gault formula
* Serum lipase =< 2 x ULN
* Serum amylase =< 2 x ULN
* International normalized ratio (INR) =< 1.5; (anticoagulation is allowed if target INR =< 1.5 on a stable dose of warfarin or on a stable dose of low molecular weight [LMW] heparin for > 2 weeks at the first dose of study agent)
* If urinalysis shows proteinuria, 24 hour urine collection is to be performed and the 24 hour urine protein is to be < 2 grams to be eligible
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Ability to understand and willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study specific procedures
* Patient must consent to the use of their archival tumor tissue for protocol use if available

Exclusion Criteria:

* Arms 2, 2E, 3, 3E: patients who previously received > 2 lines of systemic chemotherapy for advanced or metastatic disease
* Previous pelvic radiation affecting >= 25% of the bone marrow; patients who received whole pelvic radiation are excluded
* Patients who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosourea, mitomycin-C, targeted therapy and radiation) =< 4 weeks prior to starting study drug
* Patients who have received the last administration of nitrosourea or mitomycin-C =< 6 weeks prior to starting study drug
* Patients who have had radiotherapy =< 4 weeks prior to starting study drug, or =< 2 weeks prior to starting study drug in the case of localized radiotherapy (e.g., for analgesic purpose or for lytic lesions at risk of fracture)
* Patients who have received targeted therapy (e.g., sunitinib, sorafenib, pazopanib), except ALK inhibitors, =< 2 weeks prior to starting study drug
* Patients who have residual toxicity(-ities) from previous anti-cancer treatment(s) that is/are clinically significant or > grade 1 are excluded; those whose toxicity(-ities) improved to grade 1 or better will be eligible
* The patient is less than 5 half-lives from prior ALK inhibitor or targeted therapy (for adequate wash-out) without recovery from treatment toxicities to < grade 1 or to their pre-treatment levels
* Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention)
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury =< 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device =< 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Known hypersensitivity or infusion reaction to cisplatin and gemcitabine
* Patients with known hypersensitivity to any of the excipients of ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate)
* Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with ceritinib and for the duration of participation:

  * Medication with a known risk of prolonging the QT interval or inducing torsades de pointes
  * Strong inhibitors or strong inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)/5
  * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) and/or cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9)
  * Therapeutic doses (defined as doses need to achieve target INR > 1.5) of warfarin sodium (Coumadin) or any other Coumadin-derived anti-coagulant; anticoagulants not derived from warfarin are allowed (e.g., dabigatran, rivaroxaban, apixaban)
  * Unstable or increasing doses of corticosteroids
  * Enzyme-inducing anticonvulsive agents
  * Herbal supplements
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study; impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * Unstable angina within 6 months prior to screening
  * Myocardial infarction within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III - IV)
  * Uncontrolled hypertension defined by a systolic blood pressure (SBP) >= 160 mm Hg and/or diastolic blood pressure (DBP) >= 100 mm Hg, with or without antihypertensive medication
  * Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
  * Ventricular arrhythmias; supraventricular and nodal arrhythmias not controlled with medication
  * Other cardiac arrhythmia not controlled with medication
  * Corrected QT (QTc) > 450 msec using Fridericia correction on the screening electrocardiogram (ECG)
* Any active gastrointestinal (GI) impairment which, in the opinion of the investigator, would impair or alter the absorption of ceritinib (e.g., ulcerative colitis, or Crohn's disease)
* Ongoing GI adverse events > grade 2 (e.g., nausea, vomiting, or diarrhea) at the start of the study
* History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the investigator, would impair study compliance
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Pregnant or breast-feeding women
* Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test =< 3 days prior to starting study treatment
* Women of child-bearing potential, who are biologically able to conceive, not employing 2 forms of highly effective contraception; male not using at least at least one form of highly effective contraception will be excluded; highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 3 months after the end of study treatment; oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study
* Patients with untreated brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases; patients with brain metastases that have been definitively treated and on stable or decreasing dose of steroid within 4 weeks of starting study treatment will be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2015-01-08 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
MTD and RP2D of ceritinib in combination with gemcitabine hydrochloride alone, defined as the highest dose level at which < 2 of 6 patients experience treatment-related dose limiting toxicity (DLT) (Arms 1 and 1E) | Up to day 28
  Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 4.0. The frequency of toxicities will be tabulated for the dose estimated to be the MTD.
MTD and RP2D of ceritinib in combination with gemcitabine hydrochloride and cisplatin, defined as the highest dose level at which < 2 of 6 patients experience treatment-related DLT (Arms 3 and 3E) | Up to day 28
  Graded according to NCI CTCAE v4.0. The frequency of toxicities will be tabulated for the dose estimated to be the MTD.
MTD and RP2D of ceritinib in combination with gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation, defined as the highest dose level at which < 2 of 6 patients experience treatment-related DLT (Arms 2 and 2E) | Up to day 28
  Graded according to NCI CTCAE v4.0. The frequency of toxicities will be tabulated for the dose estimated to be the MTD.

SECONDARY OUTCOMES:
Incidence of adverse events of ceritinib in combination with gemcitabine hydrochloride based chemotherapy in advanced solid malignancies according to NCI CTCAE v4.0 | Up to 4 weeks after end of treatment
  Overall safety profile characterized by type, frequency, severity, timing, seriousness and relationship to study treatment. The frequency of toxicities will be tabulated by grade across all dose levels and cycles.
Pharmacokinetic parameters of ceritinib and gemcitabine hydrochloride when administered in combination in patients with advanced solid tumors (Arms 1 and 1E) | Pre-dose, 0.5, 1-2, 4-5, 6-8, and 24 hours (day 1 of courses 1-2), pre-dose on day 15 of course 1 (ceritinib); prior to end of infusion, 0.5, 1-2, and 4-6 hours post-end of infusion (day 1 of courses 1-2) (gemcitabine hydrochloride)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under the curve (AUC) or clearance (CL) of ceritinib in combination with gemcitabine hydrochloride. The effects of the cytotoxics on ceritinib pharmacokinetic will be evaluated by the model, along with other patient factors that may explain the interpatient variability in pharmacokinetics, including AUC and observed maximum concentration (Cmax).
Pharmacokinetic parameters of ceritinib, gemcitabine hydrochloride, and paclitaxel albumin-stabilized nanoparticle formulation when administered in combination in patients with advanced solid tumors (Arms 2 and 2E) | Pre-dose, 0.5, 1-2, 4-5, 6-8, and 24 hours (day 1 of courses 1-2), pre-dose on day 15 of course 1 (ceritinib); prior to end of infusion, 0.5, 1-2, and 4-6 hours post-end of infusion (day 1 of courses 1-2) (gemcitabine hydrochloride and nab-paclitaxel)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual AUCs or CL of ceritinib in combination with gemcitabine hydrochloride and nab-paclitaxel. The effects of the cytotoxics on ceritinib pharmacokinetic will be evaluated by the model, along with other patient factors that may explain the interpatient variability in pharmacokinetics, including AUC and observed Cmax.
Pharmacokinetic parameters of paclitaxel albumin-stabilized nanoparticle formulation, and cisplatin when administered in combination in patients with advanced solid tumors (Arms 3 and 3E) | Pre-dose, 0.5, 1-2, 4-5, 6-8, and 24 hours (day 1 of courses 1-2), pre-dose on day 15 of course 1 (ceritinib); prior to end of infusion, 0.5, 1-2, and 4-6 hours post-end of infusion (day 1 of courses 1-2) (gemcitabine hydrochloride and cisplatin)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual AUCs or CL of ceritinib in combination with gemcitabine hydrochloride and cisplatin. The effects of the cytotoxics on ceritinib pharmacokinetic will be evaluated by the model, along with other patient factors that may explain the interpatient variability in pharmacokinetics, including AUC and observed Cmax.
Progression free survival | Up to 4 weeks after end of treatment
Response rate as assessed by the RECIST 1.1 | Up to 4 weeks after end of treatment
  Objective tumor response will be tabulated overall (and by dose level if appropriate).

OTHER OUTCOMES:
Levels of serum and tumor biomarkers | Up to 4 weeks after end of treatment
  The relationship between ALK positivity and antitumor effects will be analyzed descriptively and simple statistics if need to.

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States